CLINICAL TRIAL: NCT02702323
Title: Treatment Patients With Pulmonary Metastasis of Liver Cancer With Apatinib Combination With TACE: a Clinical Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); The Central Hospital of Lishui City (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Ningbo No.2 Hospital (Other)
Responsible Party: Principal Investigator, guoliang shao, Vice President, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-H302
Record Dates: First submitted 2016-02-21; First posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma; Pulmonary Metastasis
Keywords: hepatocellular carcinoma; pulmonary metastasis; Apatinib; efficacy; safety
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apatinib & TACE (Experimental): Apatinib 500mg tablet by mouth per day, until disease progression, combined with TACE therapy one times every 4-6 weeks.
  Interventions: Drug: Apatinib; Procedure: TACE
- TACE (Active Comparator): TACE therapy one times every 4-6 weeks.
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: Apatinib — apatinib 500mg/day for 6 weeks began taking 4-7 days after TACE
  Arms: Apatinib & TACE
Procedure: TACE — one times every 4-6 weeks.
  Other Names: transcatheter arterial chemoembolization

SUMMARY:
This study mainly evaluate the clinical effect of Apatinib in the treatment of patients with pulmonary metastasis of hepatocellular carcinoma.Half of participants will receive Apatinib and transcatheter arterial chemoembolization (TACE) therapy in combination,while the other half will receive TACE therapy alone.

DETAILED DESCRIPTION:
Apatinib is a VEGFR targeting tyrosine kinase inhibitor, which has preliminary demonstrated the efficacy and safety in treatment of advanced hepatocellular carcinoma by phase II stage research. Pulmonary metastasis of hepatocellular cancer is one of the difficulties in clinical practice,because it's not sensitive to systemic chemotherapy.This phase Ⅲ study aims to evaluates the efficacy and safety of the Apatinib in the treatment of advanced hepatocellular cancer with pulmonary metastasis.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of hepatocellular carcinoma
* refused to sorafenib treatment
* have at least one measurable pulmonary lesions
* expected survival time ≥ 12 weeks

Exclusion Criteria:

* within four weeks before the study received radiotherapy or chemotherapy
* With a variety of factors influencing oral drugs taking and absorption (such as unable to swallow, chronic diarrhea and intestinal obstruction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival | Change from Baseline mRECIST at 12 months was assessed every 4 weeks up to 48 weeks. Data collection is from date of randomization until the date of first documented progression assessed up to 12 months.
  PFS is defined as the months that from the anticipation of the clinical-trial to the progress of hepatocellular cancer

SECONDARY OUTCOMES:
overall survival | Survival assessed every 4 weeks up to 24 months following objective disease progression. Data collection is from date of randomization until the date of death from any cause, assessed up to 48 months.
  OS is defined as the months that from the anticipation of the clinical-trial to the death of patients.
Objective response rate | 1 month post intervention
  Time to progress of lung lesions which was confirmed by CT/MRI
The Quality of Life | 0 to 24 months post intervention
Toxicity as measured by CTCAE V4.0 | 0 to 24 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: guoliang shao, phD, Study Chair — Zhejiang Cancer Hospital